CLINICAL TRIAL: NCT06863129
Title: Proximal FEmur Reconstruction or Internal Fixation fOR Metastases (PERFORM) Randomized Controlled Trial
Brief Title: Proximal FEmur Reconstruction or Internal Fixation fOR Metastases (PERFORM) Trial
Acronym: PERFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Ghert, MD (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor-Investigator, Michelle Ghert, MD, Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GHRT03
Record Dates: First submitted 2025-02-04; First posted 2025-03-07 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Bone Disease
MeSH Terms: conditions — Bone Diseases | interventions — Fracture Fixation, Internal; Plastic Surgery Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection and Reconstruction (Experimental): If a participant is randomized to the Resection and Reconstruction treatment arm, a proximal femoral resection or hip arthroplasty will be carried out as per standard surgical practice. The type of endoprosthesis used for reconstruction will be at the treating surgeon's discretion. Acetabular reconstruction (if any), the surgical approach, and the intra-operative use of cement and other adjuvants for disease control will also be at the discretion of the treating surgeon.
  Interventions: Procedure: Resection and reconstruction
- Internal Fixation (Active Comparator): If the participant is randomized to the Internal Fixation treatment arm, the surgery will involve the stabilization of the remaining bone with either an intramedullary nail, plate or screw fixation. All standard surgical principles of stable internal fixation will be followed. The type of fixation, the surgical approach, and the intra-operative use of cement and other adjuvants for disease control will be at the treating surgeon's discretion.
  Interventions: Procedure: Internal Fixation

INTERVENTIONS:
Procedure: Internal Fixation — Internal Fixation
  Arms: Internal Fixation
Procedure: Resection and reconstruction — Resection and reconstruction
  Arms: Resection and Reconstruction

SUMMARY:
The goal of this clinical trial is to find out if removing and replacing part of the hip bone works better than using metal hardware to stabilize the bone in patients whose cancer has spread to the hip. The main questions are:

1. Does removing and replacing part of the bone work better than just stabilizing it with metal hardware?
2. Does removing and replacing the bone help reduce problems like cancer coming back or the metal hardware breaking?

Researchers will compare two treatments: using metal rods and plates to stabilize the bone (internal fixation) versus removing part of the bone and possibly replacing the hip joint (resection and reconstruction) to see if the second option causes fewer problems.

Participants will:

* Be randomly assigned to one of two groups (internal fixation or resection and reconstruction).
* Have one of the two surgeries based on which group they're in.
* Go to follow-up appointments with the study doctor at 2 weeks, 6 weeks, 4 months, 6 months, 9 months, and 12 months after surgery.

DETAILED DESCRIPTION:
The Proximal FEmur Resection or Internal Fixation fOR Metastases (PERFORM) trial is a multi-centre randomized controlled trial that aims to test a paradigm shift in the oncological surgical management of patients with metastatic bone disease (MBD) of the proximal femur. The PERFORM trial will aim to determine if resection and endoprosthetic reconstruction improves patient-important outcomes compared to internal fixation in patients with MBD of the proximal femur.

MBD afflicts the majority of patients with advanced stage carcinomas and is the most common oncologic disease of the skeleton. The proximal femur is the most commonly affected location in the appendicular skeleton and is a source of significant morbidity affecting patient mobility and quality of life.

Stabilization of an impending or actual fracture of the proximal femur resulting from MBD has historically been achieved with internal fixation using intramedullary nails, plates and screws. This approach is meant to provide enough stability to ambulate without pain for the remainder of the cancer patient's life. However, many patients with metastatic cancer are experiencing longer life spans due to advances in systemic treatment options. Therefore, the traditional methods of stabilizing bones in the setting of MBD may no longer be meeting the standard of outcomes required for patients who can now live for years with their disease. Internal fixation, which is by nature a palliative surgery, results in disease relapse in nearly 20% of patients, most often due to local MBD recurrence. Alternatively, complete resection of the affected bone followed by reconstruction with an endoprosthesis, although more invasive and conferring higher surgical risks than an internal fixation procedure, reduces the risk of cancer recurrence at the surgical site to approximately 3%, thereby avoiding the deleterious effects on patient function and quality of life. However, the evidence supporting the use of resection and endoprosthetic reconstruction of the proximal femur, although promising, is retrospective and methodologically weak, resulting in a gap in the necessary evidence to change practice.

The PERFORM trial will aim to determine if resection and endoprosthetic reconstruction improves patient-important outcomes compared to internal fixation in patients with MBD of the proximal femur.

THe Methods Centre and proposed clinical sites collectively possess the methodological, logistical and clinical expertise required to successfully carry out the PERFORM trial. Ultimately, this trial has the potential to effect significant changes in orthopaedic oncology clinical practice and improve the oncologic, functional, and quality of life outcomes of patients with cancers that have metastasized to their proximal femur. While the introduction of a more invasive yet more durable procedure would represent a paradigm shift in the approach to this patient population, the challenge investigators confront is to support this practice change with high-quality, concrete evidence.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 6 months
* Lesions in the proximal femur (femoral neck, intertrochanteric region, subtrochanteric region, and combinations thereof)
* Low or intermediate risk for perioperative morbidity and/or mortality
* No more than 75% and no less than 25% bone loss
* Mutual (patient and physician) decision to perform surgical management of an impending or realized pathologic fracture due to MBD of the proximal has been made.

Exclusion Criteria:

* Lesions isolated to the femoral neck
* Lesion with any femoral head involvement
* High risk for perioperative morbidity and/or mortality
* Multidisciplinary decision that resection of the entire lesion would be indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 12 months | From enrollment to one year follow-up post surgery.
  Collected through case report forms via electronic medical records and patient/ caregiver self-reported.
Physical function | From enrollment to one year follow-up post surgery.
  Patient-Reported Outcomes Measurement Information System (PROMIS®) Global Physical Function score: To what extent are you able to carry out your everyday physical activities such as walking, climbing stairs, carrying groceries, or moving a chair? Answer options include: Completely (best outcome); Mostly; Moderately; A little; Not at all (worst outcome)
Number of days at home | From enrollment to one year follow-up post surgery.
  Patient self- reported via patient diary.

SECONDARY OUTCOMES:
Quality of life- PROMIS-PROPr (PROMIS-Preference) health utility score | From enrollment to one year follow-up post surgery.
  PROMIS-PROPr (PROMIS-Preference) utility score - encompassing mental and physical health, and quality of life. The PROMIS-PROPr combines scores from seven PROMIS domains into a single preference-based score (also called a health utility score), which captures the preferences of the general adult population. The total number of items that the patient answers are 31. This instrument gives four different scores: health utility score, domain level scores (one for each of the following domains: physical function, anxiety, depression, fatigue, sleep disturbance, social roles and activities, pain interference, cognition, and pain intensity), physical component score, and a mental component score. Answer options include: Not at all (1); A little bit (2); Somewhat (3); Quite a bit (4); Very much (5).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ghert, MD, Principal Investigator — McMaster University
Locations (6):
- United States (3):
  - Parkview Packnett Family Cancer Institute, Fort Wayne, Indiana
  - Good Samaritan Regional Medical Center, Corvallis, Oregon
  - Oregon Health and Science University Hospital, Portland, Oregon
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- AOU Città della Salute e della Scienza CTO hospital, Torino, To, Italy

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be shared with other researchers via the study website.
Supporting Information: Study Protocol
Time Frame: Throughout study period.
Access Criteria: Publicly available.
URL: https://www.performtrial.com/

REFERENCES:
- [Background] Axelrod D, Gazendam AM, Ghert M. The Surgical Management of Proximal Femoral Metastases: A Narrative Review. Curr Oncol. 2021 Sep 28;28(5):3748-3757. doi: 10.3390/curroncol28050320. PMID 34677238

DOCUMENTS (1):
  • Study Protocol (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT06863129/Prot_000.pdf